CLINICAL TRIAL: NCT04885218
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of SHR-1209 Combined With Lipid-lowering Agents in the Stable Treatment of Patients With Non-familial Hypercholesterolemia and Mixed Hyperlipidemia .
Brief Title: Efficacy and Safety of SHR-1209 Combined With Lipid-lowering Agents in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1209-302
Record Dates: First submitted 2021-04-30; First posted 2021-05-13 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Non-familial Hypercholesterolemia; Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: SHR-1209 combined with lipid-lowering agents
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1：SHR-1209 / placebo (Experimental)
  Interventions: Drug: SHR-1209 ;placebo
- Cohort 2：SHR-1209 /placebo (Experimental)
  Interventions: Drug: SHR-1209 ;placebo
- Cohort 3：SHR-1209 / placebo (Experimental)
  Interventions: Drug: SHR-1209 ;placebo

INTERVENTIONS:
Drug: SHR-1209 ;placebo — SHR-1209 and placebo 150 mg subcutaneous injection once every 4 weeks for 48 weeks
  Arms: Cohort 1：SHR-1209 / placebo
Drug: SHR-1209 ;placebo — SHR-1209 and placebo 300 mg subcutaneous injection once every 8 weeks for 48 weeks
  Arms: Cohort 2：SHR-1209 /placebo
Drug: SHR-1209 ;placebo — SHR-1209 and placebo 450 mg subcutaneous injection once every 12 weeks for 48 weeks
  Arms: Cohort 3：SHR-1209 / placebo

SUMMARY:
To evaluate the efficacy, safety, pharmacokinetics and immunogenicity of SHR-1209 subcutaneous administration in patients with non-familial hypercholesterolemia and mixed hyperlipidemia after lipid-lowering therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 on the date of signing the informed consent, male or female;
2. The report of LDL-C should be higher than the ideal lipid-lowering target according to ASCVD history;
3. Fasting triglycerides less than equal to 5.6 mmol/L；
4. Understand the study procedures and methods, volunteer to participate in the study, and sign the informed consent.

Exclusion Criteria:

1. Have the following diseases or treatment history : (1) Have known allergic reaction to experimental drugs, or have severe allergic reaction to other antibody drugs;(2) previous diagnosis of familial hypercholesterolemia according to Simon Broome Criteria;(3) cardiac function as defined by the New York Heart Association (NYHA) grade III-IV at screening or randomization or latest detected LVEF<30%;(4) CVD events within 3 months; (5) uncontrolled hypertension; (6) prior exposure to recaticimab or other PCSK9 inhibitors; (7) inadequate organ functions.
2. Any of the laboratory indicators met the following criteria at screening or at randomization :(1) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 3 times the upper limit of normal (ULN), or total bilirubin exceeding 2 times the upper limit of normal (ULN);(2) Creatine kinase (CK) exceeds 3 times the upper limit of normal value (ULN);
3. General conditions :(1) the investigator judged that subcutaneous injection was not appropriate;(2) Fertile female subjects who did not use contraception within 4 weeks before screening; Or male or female subjects who do not agree to use high-efficiency contraceptives during the trial and for 24 weeks after the last dosing;(3) Women who are pregnant or lactating.
4. The Investigator determines that the subjects have poor compliance or have any factors that may prevent them from participating in the study, including, but not limited to, the study placing the subjects at unacceptable risk or possibly interfering with the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Percentage change in LDL-C relative to baseline | at 24 weeks of treatment

SECONDARY OUTCOMES:
The value of change in LDL-C relative to baseline | at 24 weeks of treatment
Percentage change in LDL-C relative to baseline | at 48 weeks of treatment;
The value of change in LDL-C relative to baseline , | at 48 weeks of treatment;
Percentage change in non-HDL-C relative to baseline | at 24 weeks of treatment;
Percentage change in non-HDL-C relative to baseline | at 48 weeks of treatment;
Percentage change in ApoB relative to baseline | at 24 weeks of treatment;
Percentage change in ApoB relative to baseline | at 48 weeks of treatment;
Percentage change in TC/HDL-C relative to baseline | at 24 weeks of treatment;
Percentage change in TC/HDL-C relative to baseline, | at 48 weeks of treatment
Percentage change in ApoB/ApoA1 relative to baseline, | at 24 weeks of treatment;
Percentage change in ApoB/ApoA1 relative to baseline, | at 48 weeks of treatment;
Percentage change in LP (a) relative to baseline, | at 24 weeks of treatment;
Percentage change in LP (a) relative to baseline, | at 48 weeks of treatment;
Percentage change in TG relative to baseline | at 24 weeks of treatment
Percentage change in TG relative to baseline | at 48 weeks of treatment;
Percentage of patients who achieved LDL-C goal according to presence of ASCVD at baseline, | at 48 weeks of treatment;
Percentage of patients who achieved LDL-C goal according to presence of ASCVD at baseline, | at 48 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053